CLINICAL TRIAL: NCT04774419
Title: Adjuvant Checkpoint Blockade Plus Radiation In Locally Advanced, Mismatch Repair Deficient/Microsatellite Instability-High (MMR-D/MSI-H) Endometrial Cancer
Brief Title: Radiation and TSR-042 (Dostarlimab) in People With Endometrial Cancer After They Receive Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-491
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Dostarlimab; Radiation; 20-491
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Radiotherapy, Intensity-Modulated; dostarlimab

STUDY DESIGN:
Intervention Model Description: Phase II stud y Adjuvant Checkpoint Blockade Plus Radiation in Locally Advanced, Mismatch Repair Deficient/Microsatellite Instability-High (MMR-D/MSIH) Endometrial Cancer with safety run-in of adjuvant checkpoint blockade with radiation in women with Stage III-IVA, dMMR/MSI-H endometrial cancer
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiation and Dostarlimab (THIS ARM IS COMPLETED) (Experimental): Patients will undergo standard intensity modulated radiation therapy (IMRT) to the pelvic nodes and vaginal cuff (total dose of 45-50.4Gy at 1.8 Gy per fraction) for 5-6 weeks and receive IV Dostarlimab every 3 weeks for 4 cycles followed by 1 dose of 1000mg (C5). Patients will receive a maximum of 5 cycles of Dostarlimab.
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT); Drug: Dostarlimab
- Hypofractionated IMRT and Dostarlimab (Experimental): Treatment will consist of short-course, hypofractionated IMRT to deliver 25 Gy to the vaginal cuff and pelvic lymph nodes in 5 daily fractions over one week. Participants will receive TSR-042 500mg every 3 weeks over 30 minutes for 4 cycles, followed by 1 dose of 1000mg for cycle 5. For this group, in those patients who have delays in C2 of dostarlimab and/or are unable to receive the 2nd dose of dostarlimab, hypofractionated radiation may proceed independently per discretion of treating investigator in consultation with study PI. Continuation of radiation therapy will be at the discretion of the radiation oncologist in discussion with study PI/co-PIs, and can be initiated/continued independent of dostarlimab dosing. Follow-up must continue regardless of radiation treatment received.
  Interventions: Drug: Dostarlimab; Radiation: Hypofractionated IMRT

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy (IMRT) — To the pelvic nodes and vaginal cuff (total dose of 45-50.4Gy at 1.8 Gy per fraction) for 5-6 weeks.
  Arms: Radiation and Dostarlimab (THIS ARM IS COMPLETED)
Drug: Dostarlimab — IV Dostarlimab every 3 weeks for 4 cycles followed by 1 dose of 1000mg (C5). Patients will receive a maximum of 5 cycles of Dostarlimab.
  Other Names: TSR-042
Radiation: Hypofractionated IMRT — Treatment will consist of short-course, hypofractionated IMRT to deliver 25 Gy to the vaginal cuff and pelvic lymph nodes in 5 daily fractions over one week.
  Arms: Hypofractionated IMRT and Dostarlimab

SUMMARY:
This study will test whether the combination of radiation and Dostarlimab is an effective treatment for women with MMR-D/MSI-H endometrial cancer who have recently undergone surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* ECOG performance status 0-1
* Endometrial cancer: all histologies (submission of pathology report is required for all patients who underwent surgery outside of MSK)
* MMR-D or MSI-H or POLE-mutated (submission of report[s] required for. patients who underwent testing outside of MSK POLE-mutated endometrial cancers will be included regardless of MMR/MSI status and limited to up to 3 patients per group.

  * Patients with hypermethylation of MMR gene promoters (MLH1, MSH2, MSH6 or PMS2) will be included
  * POLE-mutated endometrial cancers will be included
* Must have undergone a complete surgical staging and have stage III/IVA disease.

  * Patients with measurable disease (RECIST 1.1) after surgery are NOT eligible.
  * PatienSurgery completed between 3 weeks and 12 weeks (inclusive) before cycle 1 day 1 of therapy, and must have adequately recovered from surgery and any complications of surgery.ts with isolated tumor cells in lymph nodes found on surgery will be counted as clinical stage III disease
* Surgery completed between 3 weeks and 12 weeks (inclusive) before cycle 1 day 1 of therapy, and must have adequately recovered from surgery and any complications of surgery.
* Has a negative serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential, and agrees use an adequate method of contraception from screening through 150 days after the last dose of study treatment, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  °≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use an adequate birth control method throughout the study, starting with the screening visit through 150 days after the last dose of study treatment. See list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not breastfeed during the study or for 150 days after the last dose of study treatment.
* Demonstrate adequate organ function as defined below. All screening labs should be performed within 14 days of treatment initiation.

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL
  * Creatinine Clearance GFR ≥ 45
  * Serum total bilirubin ≤ 1.5 X ULN (patients with known Gilbert's disease Serum total bilirubin who have bilirubin level ≤ 3 x ULN may be enrolled)
  * AST and ALT 3 ULN OR ≤ 5 X ULN for subjects with liver metastases
  * TSH within normal limits. If TSH is not within normal range despite no symptoms of thyroid dysfunction, normal free T4 level is required.

Exclusion Criteria:

* Has had prior chemotherapy, targeted therapy, or investigational therapy for endometrial cancer.

  °Patients who have received prior chemotherapy, targeted therapy, or other investigational therapies for other cancers and are in remission/cured may be included at the discretion of the treating investigator in consultation with the study PI.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 agent for endometrial cancer.
* Unfit for Radiation Therapy due to the following:

  * Has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
  * Patients with a prior history of pelvic radiation
  * Patients with a prior known history or current diagnosis of a vesicovaginal, enterovaginal, or colovaginal fistula.
  * Any hematological abnormality or disorder that would be a contraindication to radiation per the treating physician.
* Hypersensitivity to Dostarlimab or any of its excipients
* Patients with diagnosis of immunodeficiency or patients receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone containing antiemetic regimen or steroids as CT scan contrast premedication) may be enrolled.

  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
  * Total systemic steroid dose cannot exceed an equivalent of 10mg of prednisone daily and dose must be stable for at least 4 weeks prior to initiating protocol therapy
* Has active TB (Bacillus tuberculosis)
* Has evidence of active, non-infectious pneumonitis.
* Has history of interstitial lung disease
* Has an active infection requiring systemic therapy with intravenous antibiotics
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, and superior vena cava syndrome.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis) within the past 3 years prior to the start of treatment or patients requiring immunosuppressive therapy for the autoimmune disease. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Subjects with psoriasis not requiring systemic treatment.
* Subjects with history of immune-related hyperthyroidism with total thyroidectomy currently in remission
* Select situations after approval of study PI
* Known HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Has received a live vaccine within 30 days of planned start of study therapy.

  °Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Is unwilling to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study. The use of LAR for cognitively impaired patients is not permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer
Enrollment: 62 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) (Safety Run-in only) | up to 8 weeks
  6-18 patients will be enrolled during a safety run-in period to assess toxicities. (NCI Common Terminology Criteria for Adverse Events version 5.0)
Progression-free (PFS) | 2 years
  PFS will be defined as the number of days from the date of the first dose of drug to the date of an event of disease progression/recurrence, according to RECIST criteria version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activites), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm